CLINICAL TRIAL: NCT02582320
Title: A Retrospective Study to Evaluate the Clinical-Biologic Characteristics and Outcome of Patients Treated in Italy According to the Ibrutinib-Named Patient Program for Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: Clinical-biological Characteristics and Outcome of Chronic Lymphocytic Leukemia Under Ibrutinib-named Patient Program
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: LLC1415
Record Dates: First submitted 2015-10-15; First posted 2015-10-21 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study patients: Patients with Relapsed or refractory CLL or 17p deleted CLL fulfilling the eligibility criteria required by the Named Patient Program (NPP) who received at least 1 dose of Ibrutinib 420 mg daily before November, 30th 2014.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — A longitudinal survey will be carried out by collecting data of patients who received at least 1 dose of Ibrutinib. All patients will be observed for at least 12 months from the treatment start.

SUMMARY:
This is a retrospective observational study aimed at describing the characteristics and outcome of CLL patients included in the NPP in Italy in a period of time ranging from the start of the NPP until November, 30th 2014. A longitudinal survey will be carried out by collecting data of patients who received at least 1 dose of Ibrutinib. All patients will be observed for at least 12 months from the treatment start.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most common leukemia in adults. The disease is characterized by the progressive accumulation of phenotypically mature malignant B lymphocytes, primarily in the peripheral blood, bone marrow, and lymph nodes. Over the last 10-15 years several biological prognostic markers have been identified, starting from the immunoglobulin gene mutational analysis to CD38, ZAP70, CD49d expression, and many others. The very recent discovery of several new genes that carry point mutations in CLL, including NOTCH1, SF3B1 and BIRC3, has added more markers that seem to correlate with resistance to treatment and with transformation into Richter syndrome. A large number of chemoimmunotherapy regimens are currently considered for the treatment of CLL patients.

NPP program The Named Patient Program (NPP) is a program intended to provide early access to ibrutinib in Italy. This program is specifically for patients who have relapsed or refractory chronic lymphocytic leukaemia (CLL)/small lymphocytic lymphoma (SLL), mantle cell lymphoma.

Rationale In patients with CLL Ibrutinib, given as single agent has shown marked activity and a good safety profile. Data from patients treated with ibrutinib outside a controlled clinical trial within a National Patient Program (NPP) could give additional information about the clinical use, treatment duration, efficacy, and toxicity of ibrutinib given to CLL patients in a real life context.

ELIGIBILITY:
NPP Inclusion Criteria:

1. Patients ≥18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
3. A minimum of one prior line of systemic chemotherapy, chemo-immunotherapy, or an alemtuzumab-based regimen, consisting of at least two cycles of therapy.
4. Relapsed or refractory CLL with one or more of the following criteria:

   * Presence of deletion of the short-arm of chromosome 17 (ie 17p deletion).
   * Relapsed: Failed two or more previous treatments, at least one with a purine analogue such as fludarabine.
   * Relapsed: Progression-free interval of less than 24 months from completing treatment with a nucleoside analogue, or bendamustine-containing regimen in combination with an anti-CD20 monoclonal antibody such as rituximab.
   * Refractory: Failure to respond to a prior chemotherapy-based treatment, stable disease, or disease progression while on treatment.
5. Patient has active CLL requiring treatment as defined by the IWCLL 2008 criteria. A minimum of one of the following criteria is required:

   * Evidence of progressive marrow failure, as manifested by the development of, or worsening of, anemia or thrombocytopenia.
   * Massive (at least 6 cm below the left costal margin), progressive, or symptomatic splenomegaly.

     c. Massive nodes (at least 10 cm in longest diameter), progressive, or symptomatic lymphadenopathy.
   * Progressive lymphocytosis with an increase of more than 50% over a 2-month period or a lymphocyte doubling time of less than 6 months (which may be extrapolated). For patients with initial blood lymphocyte counts of less than 30 x 109/L (30,000/mL), lymphocyte doubling time should not be used as a single parameter to define indication for treatment. Factors contributing to lymphocytosis or lymphadenopathy other than CLL (e.g., infections) should be excluded.
   * Constitutional symptoms, defined as 1 or more of the following disease-related symptoms or signs:

     i. Unintentional weight loss >10% within the previous 6 months prior to screening.

   ii. Significant fatigue (inability to work or perform usual activities). iii. Fever higher than 38.0°C for 2 or more weeks without evidence of infection.

   iv. Night sweats for more than 1 month without evidence of infection.
6. Haematology values within the following parameters:

   * Absolute neutrophil count (ANC) of ≥0.75 x109/L independent of growth factor support.
   * Platelet count of ≥30 x109/L independent of platelet support.
7. Biochemical values within the following limits:

   * Serum creatinine ≤2 times the upper limit of normal (ULN) or estimated glomerular filtration rate (GFR [Crockcoft-Gault]) ≥30 mL/minute.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times ULN.
   * Total bilirubin ≤1.5 times ULN (unless the bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin) for whom the upper limit of serum bilirubin is 3 mg/dl.
8. No problems to swallowing regularly capsules.
9. Agreed to practice a highly effective method of birth control during and after participation in the NPP if they are of childbearing potential and sexually active.
10. Signed informed consent document (if feasible) indicating that they understand the purpose of the study, they agree to give complete access to their medical records.

NPP Exclusion criteria

1. Previous treatment with ibrutinib or participation to an ibrutinib clinical trial (ibrutinib or comparator arm).
2. Eligible to participate in a currently recruiting ibrutinib clinical trial.
3. Previously received ibrutinib as part of a clinical trial.
4. Previously received a Bruton's tyrosine kinase (BTK) inhibitor other than ibrutinib.
5. Currently enrolled in an interventional clinical trial.
6. Currently receiving chemotherapy, anticancer immunotherapy, or experimental therapy.
7. Currently recovering from acute toxicities of prior treatment for CLL.
8. Received stem cell transplantation within the past 6 months.
9. Evidence of graft-versus-host disease and/or requires immunosuppressant therapy.
10. Major surgery within the past 4 weeks or a major wound that has not fully healed.
11. History of human immunodeficiency virus (HIV) or active infection with Hepatitis C or B.
12. Ongoing uncontrolled active systemic infection.
13. Uncontrolled autoimmune haemolytic anemia (AIHA).
14. Uncontrolled idiopathic thrombocytopenic purpura (ITP).
15. Central nervous system leukemia/lymphoma or Richter's transformation.
16. Diagnosed or treated for another malignancy, other than CLL, except for:

    * Malignancy treated with curative intent and with no known active disease present for ≥3 years prior to entering this named patient program and considered to be at low risk for recurrence.
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    * Adequately treated cervical carcinoma in situ without evidence of disease.
17. Stroke within the past 6 months.
18. Intracranial haemorrhage within the past 6 months.
19. Requires anticoagulation with warfarin or equivalent vitamin K antagonist (e.g. phenprocoumon).
20. Requires treatment with a strong CYP3A inhibitor.
21. Clinically significant cardiovascular disease such as:

    * Uncontrolled or symptomatic arrhythmias.
    * Congestive heart failure.
    * Myocardial infarction within the past 6 months.
    * Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
22. Patient has any life-threatening illness, medical condition, clinically significant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with R/R CLL or 17p deleted CLL fulfilling the eligibility criteria required by the NPP who received at least 1 dose of Ibrutinib 420 mg daily before November, 30th 2014
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Number of patients who progress | At 12 months from the start of Ibrutinib

SECONDARY OUTCOMES:
Number of patients who respond to treatment | At 12 months from enrolment
  CR,PR, L-PR according to the IWCLL 2008 criteria with modification for treatment-related lymphocytosis
Treatment duration | At 12 months from enrolment
Time to next treatment in terms of number of days needed | At 12 months from treatment start
Number of patients surviving | At 12 months from treatment start
  Overall survival
Number of patients who reach normal values in the immunoglobulin levels | At 3, 6 and 12 months from treatment start
Number of patients with toxic events | At 12 months from treatment start
Number of patients who develop Richter's syndrome and secondary malignancies | At 12 months from treatment start
Number of patients who require added assistance | At 12 months from treatment start
  For example: hospitalization, emergency visits, blood product transfusions and use of hematopoietic growth factors, antibiotics.
Number of patients who fail to treatment. | At 12 months from treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Foà, Study Chair — Policlinico Umberto I, Hematology Department.
Locations (47):
- Italy (47):
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - U.O.C di Ematologia P.O. "S.Giuseppe Moscati" - 2° piano, Aversa
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Spedali Civili - Brescia - Azienda Ospedaliera - U.O. Ematologia, Brescia
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - US Dipartimentale - Centro per le malattie del sangue - Ospedale Civile - S.Giacomo, Castelfranco Veneto
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - U.O. di Medicina Interna - ASUR Marche 8 - Ospedale Civile, Civitanova Marche
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Cona
  - Unità di Ricerca e di Malattie del sangue - Ematologia San Luca Vecchio Pad. 16 - 1° Piano, Florence
  - IRCCS_AOU San Martino-IST.Clinica Ematologica, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Ospedale Niguarda " Ca Granda" - SC Ematologia Blocco SUD, Ponti Est, Scala E, 4° piano, Milan
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - Unità Trapianto di Midollo Ist. Nazionale Tumori, Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - Ospedale San Gennaro - ASL Napoli 1, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara di Sicilia
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - U.O. di Oncoematologia di Nocera Inferiore-plesso ospedaliero "A. Tortora" di Pagani del DEA Nocera-Pagani, Pagani
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Ematologia - Ospedale San Carlo, Potenza
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - U.O.C. Ematologia - IRCCS Centro oncologico della Basilicata, Rionero in Vulture
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - U.O.S.A. Ematologia ASL RMA Presidio Nuovo Regina Margherita, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Policlinico Umberto I, Hematology Department - Sapienza, Rome
  - Sezione di Ematologia Cancer Center Humanitas, Rozzano
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - A.O. Santa Maria - Terni S.C Oncoematologia, Terni
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - ULSS N.6 Osp. S. Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it